CLINICAL TRIAL: NCT04897178
Title: Use of Machine Learning Algorithms for Automated Detection of Fetal Anomalies
Brief Title: Machine Learning-based Anomaly Recognition System
Acronym: MARS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: Middle-East Obstetrics and Gynecology Graduate Education (MOGGE) Foundation (Unknown)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, Assistant lecturer, Assiut University
Other Study IDs: OBG-AI21-P1
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Fetal Anomaly
MeSH Terms: conditions — Congenital Abnormalities | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fetuses with normal anatomy: Fetuses with normal anatomy scan who demonstrate no structural abnormalities of different systems (CNS, chest and heart, abdomen, skeletal system)
  Interventions: Diagnostic Test: Ultrasound
- Fetuses with abnormal anatomy: Fetuses with abnormal anatomy scan who demonstrate any structural abnormalities that can be detected with ultrasound
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Routine 2 dimensional Ultrasound used to screen fetuses for congenital anomalies

SUMMARY:
MARS is an artificial intelligence-powered system that aims at detecting common fetal anomalies during real-time obstetrics ultrasound. The current study comprises 2 stages: (1) The stage of model creation which will include retrospective collection of images from fetal anatomy scans with known diagnoses to train these model and test their diagnostic accuracy. (2) The stage of model validation through prospective application of this model to collected videos with known normal and abnormal diagnoses

DETAILED DESCRIPTION:
Routine second trimester anomaly scan has become a routine part of antenatal care. Early detection of fetal anomalies permits patient counselling, consideration of termination if detected anomalies are considerable, and arrangement of delivery and immediate neonatal care if indicated. Furthermore, with the expanding role of fetal interventions, early detection of fetal anomalies may expand management options, some of which may lead superior outcomes compared to postnatal interventions.

However, fetal anatomy scan necessitates a particular level of training and expertise, either by sonographers or obstetricians. Unfortunately, availability of experienced personals may be globally limited. Furthermore, first trimester anatomy scan has been evolving rapidly as ultrasound machine continues to develop and clinical research yields more information on first trimester normal standards and abnormal ranges. Accordingly, first trimester scan is anticipated to be a part of routine care in the near future. Although this tool should provide substantial benefits to obstetric patients, this would require more providers with specific training, which is unlikely to be readily available.

Artificial intelligence has been incorporated in the medical field for more than 20 years. With the advancement of deep learning algorithms, deep learning has yielded exceptional accuracy in image recognition. In the last decade, deep learning exhibits high quality performance that may exceed human performance at times. One of the earliest and most prevalent applications of deep learning in medicine are radiology-related.

In the current study, the investigators will create a series of deep learning models that appraise and identify common fetal anomalies in a series of frames including recorded videos or real time ultrasound. Deep learning algorithms will be fed by labelled images of known normal and abnormal findings representing common fetal anomalies for both training and validation. These images will be collected retrospectively through medical records of contributing centers. Their diagnostic performance will be tested on retrospectively collected videos including normal and abnormal findings. In the second stage of the study, These models will be applied to prospectively collected videos of fetal anatomy scan for further validation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 18 and 45 years
* Available ultrasound image with clear findings
* postnatal confirmation of diagnosis

Exclusion Criteria:

* Absence of research authorization on medical records

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women who underwent fetal mid-trimester anatomy scan (between 18 and 22 weeks) with or without first trimester fetal anatomy scan (11-14 weeks) with documented ultrasound results and recorded images with are consistent with postnatal diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | Fetuses between 10 weeks and 32 weeks of gestation
  Diagnostic accuracy of deep learning models in identifying major fetal structural anomalies

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Aswan Faculty of Medicine, Aswān
  - Assiut Faculty of Medicine - Women Health Hospital, Asyut